CLINICAL TRIAL: NCT02301390
Title: INTERVENE: Indian Trial of Endocardial Ventricular Substrate Ablation to Prevent Recurrent VT Events
Acronym: INTERVENE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: could not meet enrollment goal
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Vivek Reddy, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B14-02-34-05
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Ventricular Tachycardia
Keywords: INTERVENE; Ventricular tachycardia; India
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Amiodarone; Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiodarone only (Active Comparator): The control group will receive amiodarone only.
  Interventions: Drug: Amiodarone
- Amiodarone + Catheter Ablation (Experimental): The experimental group will receive amiodarone plus catheter VT ablation.
  Interventions: Drug: Amiodarone; Device: Catheter Ablation

INTERVENTIONS:
Drug: Amiodarone — Amiodarone is a Class III antiarrhythmic agent.
  Other Names: Cordarone
Device: Catheter Ablation — The ablation procedure uses radiofrequency energy to destroy cardiac tissue at the origin of the arrhythmia.
  Other Names: VT catheter ablation
  Arms: Amiodarone + Catheter Ablation

SUMMARY:
This study to is being conducted in India to determine the role of catheter-based ablation for ventricular tachycardia (VT) in post- heart attack patients who meet established guidelines for implantable cardiodefibrillator (ICD) implantation, but cannot afford it. These patients would be started on chronic Amiodarone therapy, which has been shown to be effective but can often lead to multiple side effects.

Patients will therefore be randomized in an even proportion to either a) the control group, receiving chronic Amiodarone therapy, or the study group, undergoing catheter ablation of VT in addition to chronic Amiodarone therapy.

This trial will serve as a representative model for the developing world.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) accounts for approximately 50% of all cardiac death, representing an estimated annual incidence ranging from 250,000 to 350,000 cases in the United States. The pathophysiologic mechanism for sudden death in the majority of these patients is thought to be ventricular tachycardia (VT) related to coronary artery disease (CAD), which can then degenerate to ventricular fibrillation (VF). Patients who survive an initial episode of VT/VF are prone to an extremely high incidence of recurrent life-threatening events (~25% at one year). Even in patients without a history of VT/VF, the presence of CAD and left ventricular (LV) dysfunction confers a two-year mortality rate of 22%. If VT is inducible at electrophysiological testing, the two-year mortality is ~30%.

The pathogenesis of VT in the setting of CAD is reentry in the area of the scarred myocardium. After an MI, the tissue can be broadly divided into three zones: the dense scar, the surrounding live myocardial tissue, and the intervening border zone. After a myocardial infarction (MI), the "border zone" between dense scar and live tissue contains electrically-active live myocardial fibrils interspersed in areas of infarcted, fibrotic tissue-setting the stage for local reentrant circuits that result in VT.

The use of antiarrhythmic medications (AADs) to suppress the occurrence/recurrence of VT/VF in these high-risk patients has been mostly disappointing. In large clinical trials, most AADs have not only proved to be inefficacious, but to actually increase mortality. The one potential exception appears to be Amiodarone: one study suggests some mortality benefit (GESICA), while others suggest that Amiodarone provides significant antiarrhythmic benefits without a change in mortality (EMIAT, CAMIAT, SCD-HeFT). However, even the use of Amiodarone is plagued with multiple organ toxicities, ranging from pulmonary fibrosis to hepatitis, and thyroid dysfunction.

An important alternative to such questionably efficacious antiarrhythmics is the implantable cardio-defibrillator (ICD), which can accurately and effectively detect and terminate VT/VF, resulting in a significant mortality benefit in both the primary and secondary prevention of sudden cardiac death. Yet, despite these beneficial results, ICD implantation cannot be considered a cure for VT. In addition, it is common for patients to experience painful high-voltage shocks secondary to recurrent ventricular arrhythmias, or to lose consciousness prior to the delivery of therapy. Moreover, the considerable cost of ICDs severely limits their availability in the developing world-where public and/or private health insurance systems are rudimentary at best, and where the incidence of coronary artery disease is four times higher than that of the developed world-highlighting the urgency of establishing an alternative therapy for post-MI patients with ventricular arrhythmias that is both accessibly and effective.

One such option may be catheter ablation of ventricular arrhythmias. It has been well described that for hemodynamically-stable VT circuits, careful ventricular mapping to identify sites critical to the maintenance of a given circuit, followed by discrete applications of catheter-based radiofrequency (RF) energy, can effectively eliminate VT.

This strategy mocks surgical approaches that have been used extensively since the late 1970s for modification of the arrhythmogenic substrate in patients with chronic myocardial infarction. Since the location of the reentrant circuit is most often located at the junction of the normal and scarred myocardium, two effective general strategies were developed over time: a) subendocardial resection-involving surgical removal of the subendocardial layer containing the arrhythmogenic substrate in this border zone, and b) encircling endocardial ventriculotomy-consisting of the placement of a circumferential surgical lesion through the border zone and, presumably, interrupting potential VT circuits. When performed at experienced centers, the long-term freedom from malignant VT/VF after surgery is >90%. However, the significant mortality (3-14%) and morbidity associated with this invasive procedure has curtailed its use in general practice.

The less invasive, catheter approach to substrate modification relies on electroanatomical mapping systems that create a high fidelity representation of the endocardium, allowing for the reconstruction and electronic manipulation of an endocardial cast of the ventricular chamber that carefully delineates the normal and abnormal tissues. This is based on the observation that during normal sinus rhythm, there are distinguishing characteristics of the endocardial electrogram (EGM) of normal and abnormal tissue: abnormal tissue manifests lower voltage amplitude, prolonged EGM duration, and the presence of late and fractionated potentials. Marchlinski and colleagues reported in a seminal study that by using a substrate-mapping strategy, catheter-based RF ablation lesions directed in a linear fashion were effective in controlling scar-related drug-refractory unstable VT. Furthermore, using this high-density electroanatomical mapping 1) this strategy can be utilized to localize the arrhythmogenic substrate in the majority of patients with a history of myocardial infarction and sustained ventricular tachyarrhythmia's, and 2) RF ablation using an irrigated-tip ablation catheter can be effectively and safely used to modify the arrhythmogenic substrate to render VT non-inducible even in the presence of multiple VT morphologies.

The favorable results in these non-randomized reports prompted the initiation of SMASH-VT (Substrate Mapping & Ablation in Sinus Rhythm to Halt Ventricular Tachycardia Trial); a prospective randomized clinical trial to objectively assess the clinical utility of substrate ablation of scar-related VT. This trial was a randomized-controlled trial examining the role of substrate mapping and RF ablation in the primary prevention of ICD shocks in patients presenting with clinically life-threatening VT/VF. That is, patients with a history of MI, and who survive an episode of VT/VF are at high-risk for recurrent VT and thus treated with ICDs (in essence, these patients meet AVID/CIDS/CASH criteria). In normal clinical practice, these patients are not routinely treated with adjuvant medications because of their proarrhythmic potential and side effects. In addition to an ICD and routine clinical care, these patients were additionally randomized in SMASH-VT to substrate-based catheter ablation. This catheter ablation group underwent electroanatomic mapping to delineate the endocardial infarct margins (CARTO, Biosense-Webster, Inc.). Substrate modification was then performed targeting the exit sites of induced VTs and/or late potentials within the scar using standard or irrigated radiofrequency ablation catheters.

As published in late 2007 (Reddy et al, NEJM, 357:2657), the 30-day post-ablation mortality was zero, and there was no significant change in ventricular function or functional class during follow up. During an average follow-up of 22.5±5.5 months, appropriate defibrillator therapy (anti-tachycardia pacing and shocks) occurred in 21 control (33%) and 8 ablation (12%) patients (p=0.007 by the log rank test). Of these, appropriate defibrillator shocks alone occurred in 20 control (31%) and 6 ablation (9%) patients (p=0.003). Mortality was not increased in the ablation arm (control 17%, ablation 9%; p=0.29); indeed, there was a trend to decreased mortality in the ablation arm. Thus, the SMASH-VT study revealed several important points: 1) adjuvant substrate based catheter ablation is feasible in this patient population, 2) use of a saline-irrigated RF ablation catheter for this ablation strategy is safe, and 3) this strategy decreases subsequent ICD therapies in post-myocardial infarction patients receiving defibrillators for the secondary prevention of sudden death.

The favorable results of SMASH-VT, combined with considerable technical and scientific improvements in catheter ablation of scar-related VT, also raise the possibility that the therapeutic benefit of ablation may be extrapolated to similar patients in the developing world, who have had an MI and have survived a ventricular arrhythmic event, but are unable to afford an ICD. This is of particular importance because such patients are typically treated with chronic Amiodarone therapy-a strategy with an unestablished mortality benefit and significant side effects.

The investigators therefore propose a randomized clinical trial, in which India-a nation with a population of 1.2 billion-will serve as a representative model for the developing world. The study will evaluate the safety and efficacy of adjunctive catheter ablation in post-myocardial infarction patients who have additionally survived a ventricular arrhythmic event, and would be initiated on chronic Amiodarone therapy because of an inability to afford ICD therapy. Patients will therefore be randomized in an even proportion to either a) the control group, receiving chronic Amiodarone therapy, or the study group, undergoing catheter ablation of VT in addition to chronic Amiodarone therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 85 years of age
* History of a remote MI (≥1 month)
* Survival of a ventricular arrhythmic event (VT/VF) that would mandate placement of an implantable cardioverter-defibrillator (ICD) (Patients who experience a ventricular arrhythmic event (VT/VF) while already being treated with Amiodarone (100-200 mg/day) are not excluded from the study. This is permitted provided that the patient had been treated with Amiodarone for at least 2 months prior to experiencing the index VT/VF event. These patients are randomized to either a higher dose of Amiodarone (e.g., 100mg/day -> 200mg/day or 200mg/day -> 400mg/day) or a higher dose of Amiodarone plus catheter ablation.)
* Patient cannot afford an ICD and thus has been planned for treatment with Amiodarone (or an increased dose of Amiodarone)
* Ability to understand the requirements of the study
* Willingness to adhere to study restrictions and comply with all post- procedural follow-up requirements

Exclusion Criteria:

* Patients with NYHA class IV congestive heart failure
* Prior ablation for a ventricular arrhythmia
* Presence of an LV thrombus
* Contraindication to anticoagulation
* Inability to access the endocardium because of mechanical mitral and aortic valve
* Life expectance <1 year for any medical condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Calambur Narasimhan, MD, Principal Investigator — CARE Hospital
Locations (3):
- India (3):
  - CARE Institute of Medical Science, Ahmedabad
  - CARE Hospital, Hyderabad
  - Jawaharlal Institute of Postgraduate Medical Education and Research (JIPMER), Puducherry

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Amiodarone Only: Amiodarone is a Class III antiarrhythmic agent.
- Amiodarone + Catheter Ablation: Amiodarone is a Class III antiarrhythmic agent.
  Catheter VT Ablation: The ablation procedure uses radiofrequency energy to destroy cardiac tissue at the origin of the arrhythmia.
Period: Overall Study
Arm/Group | Amiodarone Only | Amiodarone + Catheter Ablation
Started | 27 | 26
Completed | 17 | 13
Not Completed | 10 | 13
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 2 | 2
Not completed — Procedure not completed | 0 | 4
Not completed — Missed multiple visits | 1 | 1
Not completed — study terminated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amiodarone Only | Amiodarone + Catheter Ablation | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (10.7) | 53.8 (10.4) | 54.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 26 | 24 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 26 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 26 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Free From All-cause Mortality, Sustained VT or Cardiac Arrest
Description: Number of participants who had no occurrences of all-cause mortality, sustained ventricular tachycardia (VT) and cardiac arrest at 24 months
Time Frame: at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone Only | Amiodarone + Catheter Ablation
Number analyzed (Participants) | 27 | 26
Participants | 16 | 21

2. Secondary Outcome: Number of Participant Who Died
Description: Number of subjects that die within 30 days or die by 24 months.
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Amiodarone Only | Amiodarone + Catheter Ablation
Number analyzed (Participants) | 27 | 26
Participants
  within 30 days | 0 | 0
  24 months | 2 | 2

3. Secondary Outcome: Ventricular Arrhythmic Events
Description: Total number of ventricular arrhythmic events, compared between the 2 treatment arms.
Time Frame: at 24 months
Measure: Number; unit: events
Arm/Group | Amiodarone Only | Amiodarone + Catheter Ablation
Number analyzed (Participants) | 27 | 26
events | 15 | 5

4. Secondary Outcome: Change in LV Ejection Fraction
Description: Change in left ventricle (LV) ejection fraction between paired measurements recorded at 24 months as compared to baseline
Time Frame: baseline and 24 months
Population: Data for only those who had two time points LV ejection fraction data
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Amiodarone Only | Amiodarone + Catheter Ablation
Number analyzed (Participants) | 14 | 8
percent | 1.85 (6.32) | 8 (.31)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Amiodarone Only | Amiodarone + Catheter Ablation
All-Cause Mortality (participants affected / at risk) | 2/27 | 2/26
Serious Adverse Events (participants affected / at risk) | 11/27 | 8/26
Other Adverse Events (participants affected / at risk) | 4/27 | 6/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amiodarone Only (N=27) | Amiodarone + Catheter Ablation (N=26)
VT recurrrence (Cardiac disorders) | 10 | 5
Bradycardia (Cardiac disorders) | 1 | 0
Heart Failure (Cardiac disorders) | 2 | 1
LV failure (Cardiac disorders) | 2 | 0
CVA (General disorders) | 0 | 1 — Cerebrovascular accident (CVA)
Motor aphasia (Nervous system disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Subclinical/Sub radiological ILD (Cardiac disorders) | 1 | 0 — Interstitial Lung Disease (ILD)
Amiodarone induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic enephalopathy (Hepatobiliary disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amiodarone Only (N=27) | Amiodarone + Catheter Ablation (N=26)
Bradycardia (Cardiac disorders) | 2 | 3
Hypothyroidism (Endocrine disorders) | 0 | 1
Transient AV block while crossing the Aortic Valve (Cardiac disorders) | 0 | 1
Chronic progressive gingivitis (General disorders) | 0 | 1
right foot injury (Musculoskeletal and connective tissue disorders) | 0 | 1
Viral Pyrexia (Infections and infestations) | 0 | 1
Frequent loose stools (Gastrointestinal disorders) | 0 | 1
Frequent loose stools (Gastrointestinal disorders) | 1 | 0
anxiety (Psychiatric disorders) | 1 | 0
Right arm ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT02301390/Prot_SAP_000.pdf